CLINICAL TRIAL: NCT02650700
Title: Spleen Radiotherapy Decreases Severe Chemotherapy Induced Thrombocytopenia (CIT) for the Multi-center Randomized Controlled Study in Advanced NSCLC
Brief Title: Spleen Radiotherapy Decreases Severe CIT in Advanced NSCLC (SPLEENIR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy director,Xinqiao Hospital of Chongqing, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-002
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Chemotherapy in Non-Small Cell Lung Cancer
Keywords: spleen radiation; IMRT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spleen radiation plus spleen radiotherapy (Experimental): Chemotherapy plus spleen radiotherapy Chemotherapy plus spleen radiotherapy are performed, simultaneously, to the subjects with advanced lung cancer who experienced chemotherapy induced thrombocytopenia (≧grade II CIT). The intervention is spleen radiotherapy.
  Interventions: Radiation: spleen radiotherapy
- chemotherapy (Other): Chemotherapy is performed to the subjects with advanced lung cancer who experienced chemotherapy induced thrombocytopenia (≧grade II CIT). When severe CIT (≧grade III) occurs, the subjects should receive chemotherapy plus spleen radiotherapy. The intervention is spleen radiotherapy.
  Interventions: Radiation: spleen radiotherapy

INTERVENTIONS:
Radiation: spleen radiotherapy — Radiation: spleen radiation In Experimental arm, combine spleen radiation with chemotherapy. In Chemotherapy alone arm, the subjects should also receive spleen radiation once there is a severe CIT (≧grade III) during chemotherapy after radomization.
  Other Names: IMRT

SUMMARY:
Chemotherapy is one of the main treatments for advanced NSCLC. However, chemotherapy induced thrombocytopenia (CIT) is one of the most important limitations for subsequent chemotherapy of cancer.

Although platelet transfusion is the gold standard to treat severe CIT, its clinical application is limited due to many disadvantages, such as short time for storage, not easy to save, the risk of infection and immunological diseases. What's more, other cytokines including IL-11 and rhTPO, are not so useful in clinical work. It is necessary to explore a new therapeutic method to treat CIT.

Researches show that spleen resection could improve the count of PLT. In this clinical trial, we design chemotherapy plus spleen radiotherapy to the subjects with advanced NSCLC, simultaneously, who underwent grade II or worse CIT. The primary endpoint is the incidence of severe CIT (≧grade III) in subsequent chemotherapy, the second endpoints are recovery time from bone marrow suppression and progression free survival, and the exploring index is the immulogical status.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced (Stage IIIA or IIIB AJCC 7) NSCLC that was histologically or cytologically inoperable
2. ECOG whole body status (performancestatus,PS) level 0 or 1
3. The estimated survival time is more than 12 weeks, 18 ~75 years old
4. Laboratory results within 2 weeks prior to radiotherapy met the following criteria: ① Neutrophil count > 1,500/ MCL Heathko-Pilot Oncology Research Fund; ② Platelet > 50,000/ MCL; ③ Total bilirubin < 1.5 times of the normal upper limit value; ④AST(SGOT)/ALT(SGPT) < 2.5 times of the normal upper limit; ⑤ Serum creatinine < 1.5 times of the normal upper limit value; ⑥ The results of coagulation function examination were within the normal range
5. Women of childbearing age must have taken reliable contraceptive measures or conducted pregnancy tests (serum or urine) within 7 days before admission, and the results are negative, and are willing to use appropriate methods of contraception during the trial period and 8 weeks after the last administration of the trial drug. For men, they must agree to use appropriate methods of contraception or surgical sterilization during the trial period and 8 weeks after the last administration of the trial drug
6. Understand and voluntarily sign written informed consent
7. The investigator judged that the patient had good compliance

Exclusion Criteria:

1. Patients with serious functional damage of important organs;
2. Patients diagnosed adequately with other malignant tumors;
3. Pregnant or lactating women;
4. Patients in an active period of acute or chronic infectious diseases;
5. Combined with the disease of connective tissue
6. Patients who are allergic to any drugs or people with allergies;
7. Patients who participate in other clinical trials concurrently;
8. Brain metastases without being controlled;
9. With immunologic thrombocytopenia；
10. Excluding thrombocytopenia caused by other reasons(Non chemotherapeutic agents, such as heparin, etc.);
11. The degree of tumor thrombus >2;
12. Patients who are considered not eligible for the trial after evaluation by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
The incidence of severe CIT afer chemotherapy | 18 weeks after randomization

SECONDARY OUTCOMES:
Recovery time after severe bone marrow suppression | 18 weeks after randomization
Progression free suvival (PFS) | Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months
Objective response rate (ORR) | Time Frame: 18 weeks after randomization